CLINICAL TRIAL: NCT02445313
Title: Measuring Geographic Atrophy in AMD Patients Using the Nidek MP-3 Microperimetry Device
Status: Completed | Type: Observational
Sponsor: Doheny Image Reading Center (Other)
Responsible Party: Sponsor
Other Study IDs: NIDEKMP3
Record Dates: First submitted 2015-05-13; First posted 2015-05-15 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Age-related Macular Degeneration (AMD)
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Normal, healthy participants
  Interventions: Device: Nidek MP-3
- AMD: Age-related Macular Degeneration participants
  Interventions: Device: Nidek MP-3

INTERVENTIONS:
Device: Nidek MP-3 — Nidek MP-3 device to be used to take images which will allow measurement of GA in patients with AMD

SUMMARY:
The investigators would like to know if different imaging devices can improve the quality of images and visualization of imaged tissues. Also, the investigators would like to find out whether these changes are useful in the diagnosis and treatment of eye diseases. Using images of previous participants will allow us to demonstrate the advancement of different technologies, as well be used to allow comparisons between current technologies.

DETAILED DESCRIPTION:
To test the quality of images from the Nidek MP-3 device and to measure Geographic Atrophy (GA) in patients with Age-related Macular Degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

* Normal, healthy participants and patients with AMD

Exclusion Criteria:

1. Those suffering from head, neck or other injury which makes them unable to position themselves in head restraint for imaging
2. Participants who are unable to maintain retinal fixation on a specified target
3. Participants unable to achieve sufficient pupil dilation and alignment stability for imaging to take place
4. Patients with media opacity which preclude high quality imaging will be excluded.
5. Exclusion criteria include vulnerable patients; patients under 18, pregnant, economically and educationally disadvantaged, decision impaired, or homeless people. We exclude pregnant women because pregnancy often can alter eye anatomy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cohort A will consist of patients with AMD, recruited by PI when they come in to the clinic, with whom we will conduct medical record review and imaging procedures, using one of the research devices.
  Cohort B will consist of control subject with no ocular problems, with whom no record review will be conducted, but imaging will be conducted with study devices.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-06; Primary Completion 2019-02-12 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
Geographic Atrophy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas Sadda, Principal Investigator — Doheny Eye Institute
Locations (1):
- Doheny Eye Centers UCLA, Pasadena, California, United States